CLINICAL TRIAL: NCT03104556
Title: Silent sTROke duriNG MitraClip Implantation - STRONG-MitraClip
Brief Title: Silent sTROke duriNG MitraClip Implantation
Acronym: STRONG
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Alexander Lauten, Prof. Dr. med. A. Lauten, Charite University, Berlin, Germany
Other Study IDs: STRONG-MitraClip 01
Record Dates: First submitted 2017-04-01; First posted 2017-04-07 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Mitral Regurgitation; Silent Stroke
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The MitraClip-procedure offers an interventional treatment for high risk patients with severe symptomatic mitral regurgitation. The number of new cerebral ischemic lesions without clinical manifestations is high. The aim of this study is to determine the frequency of cerebral embolisms and cerebral lesions during the MitraClip-procedure using transcranial doppler ultrasound and magnetic resonance imaging.

DETAILED DESCRIPTION:
Mitral regurgitation is the second most common manifestation of valvular heart disease in adults. Surgical reconstruction is considered treatment of choice. For some patients the surgical risk is to high an operation is refused. For those Patients the MitraClip system (Abbott Vascular, Menlo Park, CA, USA) offers a much less invasive treatment option. Occurrence of a stroke or transient ischemic attack (TIA) is one of the potential complications during this procedure. 1% of all patients have an acute stroke. The number of new ischemic lesions without clinical manifestations is much higher (up to 85%). The impact of these lesions on the global cognitive function is unclear. The aim of this study is to determine the frequency of cerebral embolisms related to predefined procedural intervals and postprocedural cerebral lesions using Transcranial Doppler ultrasound and magnetic resonance imaging. Furthermore we want to study the correlation between cerebral embolisms seen as high intensity signals in transcranial duplex ultrasound and cerebral lesions seen in the cMRT. The results should build a basis for further studies that want to reduce the amount of cerebral lesions.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing a MitraClip-procedure due to mitral regurgitation in the study period Written consent Procedure recommended by a Cardio-Thoracic Surgery Conference

Exclusion Criteria:

Patients who are not able to give consent Patients <18 years Participation in another interventional Trial Pregnant or lactating females Contraindication to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing the MitraClip between April 2017 December 2019 procedure due to a severe mitral regurgitation will be enrolled in our study. All patients will be assigned to either a surgical procedure or the MitraClip-procedure by an interdisciplinary heart team according to current guidelines irrespective of this study.
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2017-04-14 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2020-12-03 (Actual)

PRIMARY OUTCOMES:
Total amount of high intensity signals (HITS) during the predefined procedural intervals | during the procedure

SECONDARY OUTCOMES:
Total amount of high intensity signals and cerebral lesions related to primary and secondary mitral regurgitation | 0-72h
Localizations of cerebral lesions after MitraClip-procedure | 0-72h
Incidence of peri- and postprocedural stroke | 0-72h
Incidence of delirium after MitraClip | 0-72h

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Lauten, Prof. Dr., Study Chair — Charite Kardiologie
Locations (1):
- Charite, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Braemswig TB, Kusserow M, Bellmann B, Beckhoff F, Reinthaler M, von Rennenberg R, Erdur H, Scheitz JF, Galinovic I, Villringer K, Leistner DM, Audebert HJ, Endres M, Landmesser U, Haeusler KG, Fiebach JB, Lauten A, Rillig A, Nolte CH. New Cerebral Microbleeds After Catheter-Based Structural Heart Interventions: An Exploratory Analysis. J Am Heart Assoc. 2023 Feb 7;12(3):e8189. doi: 10.1161/JAHA.122.027284. Epub 2023 Feb 3. PMID 36734351